CLINICAL TRIAL: NCT05170646
Title: Real World Clinical and Patient-Reported Outcomes of Patients With Moderate-to-Severe Rheumatoid Arthritis Initiating Upadacitinib in the United Kingdom: A Prospective, Observational Cohort Study
Brief Title: An Observational Study to Assess the Real-World Effectiveness of Upadacitinib in Adult Participants With Rheumatoid Arthritis
Acronym: ENDEAVOUR
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-235
Record Dates: First submitted 2021-11-16; First posted 2021-12-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis (RA); Upadacitinib; RINVOQ
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants treated with upadacitinib

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease causing pain, stiffness, swelling and loss of joint function. RA can reduce the ability to perform everyday tasks. This study will assess the clinical and patient-reported outcomes with upadacitinib in adult participants with moderate-to-severe RA in a real-world setting.

Upadacitinib is an approved drug for the treatment of adults with moderately to severely active RA who have had an inadequate response or intolerance to methotrexate. Adult participants with moderate-to-severe RA will be enrolled. Around 150 participants will be enrolled in the study in multiple sites in the United Kingdom.

Participants will receive upadacitinib per their physician's usual prescription. Individual data will be collected for 6 months.

No additional study-related tests will be conducted during the routine physician visits. Only data which are routinely collected during a regular visit will be utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology (ACR) or European League Against Rheumatism (EULAR) confirmed diagnosis of rheumatoid arthritis (RA).
* Moderate RA (defined by National Institute for Health and Care Excellence [NICE] as 28-joint Disease Activity Score [DAS28] C-reactive protein [CRP] >3.2 and ≤5.1) or severe RA (defined by NICE as DAS28 CRP >5.1) at the time of enrollment.
* Prescribed upadacitinib in line with marketing authorization.
* Decision to treat with upadacitinib has been made independently and prior to enrolment in the study.
* Able to read and understand English.
* Willing and able to participate in the collection of patient-reported data via mobile app.

Exclusion Criteria:

* First dose of upadacitinib received prior to enrollment in the study (same day permitted) or more than 28 days after enrolment into the study.
* Previously received >4 biologic disease-modifying antirheumatic drugs (bDMARD) (1 switch to a biosimilar for non-clinical reasons is allowed for each bDMARD received) or any Janus kinase (JAK) inhibitor for the treatment of RA.
* In the opinion of the treating clinician, participant symptoms are predominately being driven by fibromyalgia or unrelated pain component instead of underlying inflammatory disease.
* Participation in any interventional clinical trial within the 3 months prior to initiation or at any point during the study observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Participants with moderate-to-severe rheumatoid arthritis (RA)
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving 28-Joint Disease Activity Score (DAS28) C-reactive protein (CRP) Clinical Remission | 6 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Clinical remission is defined as a DAS28 CRP <2.6.

SECONDARY OUTCOMES:
Percentage of Participants Achieving a Moderate European League Against Rheumatism (EULAR) Response | 6 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. A moderate EULAR response is defined as a DAS28 CRP >5.1 with a DAS28 CRP decrease >1.2 or DAS 28 CRP score >3.2 and ≤5.1 with DAS28 CRP decrease >0.6.
Percentage of Participants Achieving DAS28 CRP Clinical Remission | 3 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Clinical remission is defined as a DAS28 CRP <2.6.
Percentage of Participants Achieving DAS28 CRP Low Disease Activity | 3 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Low disease activity is defined as DAS28 CRP <=3.2.
Percentage of Participants Achieving DAS28 CRP Low Disease Activity | 6 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Low disease activity is defined as DAS28 CRP <=3.2.
Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Clinical Remission | 3 Months
  The CDAI is a validated measure of RA disease activity. Scores on the CDAI range from 0 (lowest disease activity) to 76 (highest disease activity). Clinical remission is defined as CDAI <=2.8.
Percentage of Participants Achieving CDAI Low Disease Activity | 3 Months
  The CDAI is a validated measure of RA disease activity. Scores on the CDAI range from 0 (lowest disease activity) to 76 (highest disease activity). Low disease activity is defined as CDAI <=10.
Percentage of Participants Achieving CDAI Clinical Remission | 6 Months
  The CDAI is a validated measure of RA disease activity. Scores on the CDAI range from 0 (lowest disease activity) to 76 (highest disease activity). Clinical remission is defined as CDAI <=2.8.
Percentage of Participants Achieving CDAI Low Disease Activity | 6 Months
  The CDAI is a validated measure of RA disease activity. Scores on the CDAI range from 0 (lowest disease activity) to 76 (highest disease activity). Low disease activity is defined as CDAI <=10.
Percentage of Participants Achieving Boolean Remission | 3 Months
  Boolean remission is achieved when all of the following conditions are satisfied: tender joint count <=1, swollen joint count <=1, CRP <=1 mg/dL, and patient global assessment <=1 (on a 0-10 scale).
Percentage of Participants Achieving Boolean Remission | 6 Months
  Boolean remission is achieved when all of the following conditions are satisfied: tender joint count <=1, swollen joint count <=1, CRP <=1 mg/dL, and patient global assessment <=1 (on a 0-10 scale).
Percentage of Participants Initiating Upadacitinib as Monotherapy | Baseline
  Percentage of participants initiating upadacitinib without conventional synthetic disease-modifying antirheumatic drugs (csDMARDs).
Percentage of Participants Initiating Upadacitinib in Combination Therapy | Baseline
  Percentage of participants initiating upadacitinib in combination therapy with csDMARDs.
Time to Discontinuation of Upadacitinib | Up to 6 Months
  Time from initiation to discontinuation of upadacitinib.
Percentage of Participants Remaining on Treatment | 6 Months
  Percentage of participants remaining on upadacitinib 6 months post initiation.
Number of Other (Not Rheumatoid Arthritis [RA]-Related) Concomitant Medications Prescribed | Baseline
  Other (not RA-related) concomitant medications include statins and other non-RA-related concomitant medications.
Number of RA-Related Concomitant Medications Prescribed | Up to 6 Months
  RA-related concomitant medications include csDMARDS, corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), other painkillers, and other RA-related concomitant medications.
Percentage of Participants Who Have Received any COVID-19 or Herpes Zoster Vaccination | Up to 6 Months
  Percentage of participants who have received any COVID-19 or Herpes Zoster vaccination and a summary of vaccination details.
Change from Baseline in Pain Visual Analogue Scale (VAS) | Up to 6 Months
  The patient's level of pain in the last 24 hours will be measured using a pain VAS. VAS scores range from 0 to 100 points with a higher score indicating more pain.
Change from Baseline in Fatigue VAS Score | Up to 6 Months
  A fatigue VAS will be used to assess the patient's level of fatigue on a weekly basis. VAS scores range from 0 to 100 points with a higher score indicating more fatigue.
Change from Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score | Up to 6 Months
  The FACIT-Fatigue Scale measures an individual's level of fatigue during their usual daily activities over the past week. on a four-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The score range for FACIT-Fatigue is between 0 and 52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life.
Change from Baseline in Patient Health Questionnaire-2 (PHQ-2) Score | Up to 6 Months
  The PHQ-2 screens for the presence of possible depression. The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past 2 weeks, scoring each component from 0 ("not at all") to 3 ("nearly every day").
Change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score | Up to 6 Months
  The HAQ-DI assesses physical function in RA. The HAQ-DI score is the average of the highest score in each of eight categories. The total score is between 0-3.0, in 0.125 increments. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment
Change from Baseline in EQ-5D-5L Score | Up to 6 Months
  The EQ-5D-5L comprises of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. In addition, a vertical VAS is used to assess patient's self-rated health status. The endpoints for the VAS are labelled 'the best health you can imagine' and 'the worst health you can imagine'. The recall period is one day.
Change from Baseline in Work Productivity and Activity Impairment Questionnaire-General Health (WPAI-GH) Score | Up to 6 Months
  The WPAI-GH measures the impact of health problems on absenteeism, presenteeism, overall work performance and non-work activities using a 0 to 10 VAS.
Percentage of Participants Achieving Minimal Clinically Important Difference (MCID) in Pain VAS | Up to 6 Months
  The patient's level of pain in the last 24 hours will be measured using a pain VAS. VAS scores range from 0 to 100 points with a higher score indicating more pain. MCID is defined as at least a 10 point difference from baseline.
Percentage of Participants Achieving MCID in Fatigue VAS Score | Up to 6 Months
  A fatigue VAS will be used to assess the patient's level of fatigue on a weekly basis. VAS scores range from 0 to 100 points with a higher score indicating more fatigue. MCID is defined as a decrease of -1.12.
Percentage of Participants Achieving MCID in FACIT-Fatigue Score | Up to 6 Months
  The FACIT-Fatigue Scale measures an individual's level of fatigue during their usual daily activities over the past week. on a four-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The score range for FACIT-Fatigue is between 0 and 52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life. MCID is defined as a 4-point increase.
Percentage of Participants Achieving MCID in PHQ-2 Score | Up to 6 Months
  The PHQ-2 screens for the presence of possible depression. The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past 2 weeks, scoring each component from 0 ("not at all") to 3 ("nearly every day"). MCID is defined as achievement of a PHQ-2 score <=2 and absence of low mood.
Percentage of Participants Achieving MCID in HAQ-DI Score | Up to 6 Months
  The HAQ-DI assesses physical function in RA. The HAQ-DI score is the average of the highest score in each of eight categories. The total score is between 0-3.0, in 0.125 increments. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment. MCID is defined as decrease of -0.22.
Time to Achieve MCID in FACIT-Fatigue Score | Up to 6 Months
  The FACIT-Fatigue Scale measures an individual's level of fatigue during their usual daily activities over the past week. on a four-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The score range for FACIT-Fatigue is between 0 and 52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life. MCID is defined as a 4-point increase.
Time to Achieve MCID in Pain VAS | Up to 6 Months
  The patient's level of pain in the last 24 hours will be measured using a pain VAS. VAS scores range from 0 to 100 points with a higher score indicating more pain. MCID is defined as at least a 10 point difference from baseline.
Time to Achieve MCID in Fatigue VAS Score | Up to 6 Months
  A fatigue VAS will be used to assess the patient's level of fatigue on a weekly basis. VAS scores range from 0 to 100 points with a higher score indicating more fatigue. MCID is defined as a decrease of -1.12.
Time to Achieve MCID in PHQ-2 Score | Up to 6 Months
  The PHQ-2 screens for the presence of possible depression. The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past 2 weeks, scoring each component from 0 ("not at all") to 3 ("nearly every day"). MCID is defined as achievement of a PHQ-2 score <=2 and absence of low mood.
Time to Achieve MCID in HAQ-DI Score | Up to 6 Months
  The HAQ-DI assesses physical function in RA. The HAQ-DI score is the average of the highest score in each of eight categories. The total score is between 0-3.0, in 0.125 increments. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment. MCID is defined as decrease of -0.22.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- United Kingdom (15):
  - University Hospitals of Morecambe Bay NHS Foundation Trust /ID# 242376, Kendal, Cumbria
  - Leicester Royal Infirmary /ID# 244674, Leicester, England
  - Medway NHS Foundation Trust /ID# 244673, Gillingham, Kent
  - Guys and St Thomas NHS Foundation Trust /ID# 251704, London, London, City of
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 251700, Norwich, Norfolk
  - Northampton General Hospital NHS Trust /ID# 251710, Northampton, Northamptonshire
  - Royal United Hospitals Bath /ID# 251707, Bath
  - Cambridge University Hospitals NHS Foundation Trust /ID# 251706, Cambridge
  - Liverpool University Hospitals NHS Foundation Trust /ID# 251701, Liverpool
  - King's College Hospital NHS Foundation Trust /ID# 251705, London
  - Western Health and Social Care Trust /ID# 251702, Londonderry
  - Luton and Dunstable Hospital NHS Foundation Trust /ID# 251699, Luton
  - Aneurin Bevan University Health Board /ID# 251703, Newport
  - The Royal Wolverhampton NHS Trust /ID# 251708, Wolverhampton
  - York and Scarborough Teaching Hospitals NHS Foundation Trust /ID# 244672, York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-235#additional-resources-section